CLINICAL TRIAL: NCT02173652
Title: Pharmacokinetics and Pharmacodynamics of Multiple 5 mg Doses of BI 1356 p.o. Given Once Daily Compared to Multiple 2.5 mg Doses Given Twice Daily in Healthy Male and Female Volunteers. A Monocentric, Open Label, Cross-over Trial
Brief Title: Pharmacokinetics and Pharmacodynamics of Multiple 5 mg Doses of BI 1356 p.o. Given Once Daily Compared to Multiple 2.5 mg Doses Given Twice Daily in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1218.45
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin

ARMS (2):
- BI 1356, high dose (Experimental): Treatment A: 7 days of BI 1356 treatment given once daily
  Interventions: Drug: BI 1356, high dose
- BI 1356, low dose (Active Comparator): Treatment B: 7 days of BI 1356 treatment given twice daily
  Interventions: Drug: BI 1356, low dose

INTERVENTIONS:
Drug: BI 1356, high dose
  Arms: BI 1356, high dose
Drug: BI 1356, low dose
  Arms: BI 1356, low dose

SUMMARY:
The objective was to investigate the influence of 2 different dosage regimens (5 mg once daily vs. 2.5 mg twice daily) on the steady-state pharmacokinetics and pharmacodynamics of orally administered BI 1356.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females and males based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age ≥18 and Age ≤65 years
* BMI ≥18.5 and BMI ≤29.9 kg/m² (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections (e.g. HIV)
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsade de pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

For male subjects:

* Not willing to use adequate contraception (condome use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, IUD (intrauterine device)) during the whole study period from the time of the first intake of study drug until one month after the last intake

For female subjects:

* Pregnancy or planning to become pregnant within 2 months of study completion
* Positive pregnancy test
* Are not willing or are unable to use a reliable method of contraception (such as implants, injectibles and combined oral contraceptives, sterilisation, IUD, double barrier method) for at least 3 months prior to participation in the trial, during and up to 2 months after completion/termination of the trial
* Chronic use of oral contraception or hormone replacement containing ethinyl estradiol as the only method of contraception
* Lactation period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
AUC0-24,ss (area under the concentration-time curve of the analyte in plasma over the time interval 0 to 24 hours at steady state) | up to 336 h after first administration of study drug

SECONDARY OUTCOMES:
Cmax,ss (concentration of the analyte in plasma at steady state after administration of the last dose at the end of the dosing interval) | up to 336 h after first administration of study drug
Cpre,N (predose concentration of the analyte in plasma immediately before administration of the Nth dose after N-1 doses were administered) | up to 336 h after first administration of study drug
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 336 h after first administration of study drug
AUCss (area under the concentration-time curve of the analyte in plasma at steady state) for several time points | up to 336 h after first administration of study drug
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) | up to 336 h after first administration of study drug
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) | up to 336 h after first administration of study drug
CLR,ss (renal clearance of the analyte at steady state determined over the dosing interval τ) | up to 336 h after first administration of study drug
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | up to 336 h after first administration of study drug
Aet1-t2 (amount of BI 1356 excreted in the urine over the time interval t1 to t2 at steady-state) | 0-12h and 12-24h after drug administration on day 7 and day 14
fet1-t2 (fraction of BI 1356 excreted in urine over the time interval form t1 to t2) | 0-12h and 12-24h after drug administration on day 7 and day 14
Number of patients with clinically relevant findings in vital signs (blood pressure (BP), pulse rate (PR)) | Baseline, up to 26 days
Number of patients with clinically relevant findings in 12-lead ECG (electrocardiogram) | Baseline, up to 26 days
Number of patients with clinically relevant findings in clinical laboratory tests | Baseline, up to 26 days
Incidence of adverse events (AEs) | up to 47 days
Assessment of tolerability on a 4-point scale by investigator | Day 7, 15 and 26
Dipeptidyl peptidase-4 (DPP-4) inhibition at steady state | up to 336 h after first administration of study drug